CLINICAL TRIAL: NCT03365076
Title: Exercise for Improving Prostate Oxygenation in Prostate Tumors (Exipox)-Study - a Pilot Study Exploring Exercise as a Way of Improving Cure With Radical Radiotherapy
Brief Title: Exercise for Improving Prostate Oxygenation in Prostate Tumors (Exipox)
Acronym: EXIPOX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow inclusion rate due to patients operated before intervention is implementable
Sponsor: University Hospital of North Norway (Other)
Collaborators: Oslo University Hospital (Other); University of Tromso (Other); Northern Health Authority (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1791
Record Dates: First submitted 2017-10-06; First posted 2017-12-07 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer; Physical Activity; Hypoxia
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity; Hypoxia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Open label randomized control trial. Randomization 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical aerobic intervention (Experimental): The exercise program will be varying between different aerobic activities indoor or outdoor as walking uphill and in stairs in intervals that will differ from session to session to build up the load and progression for these patients. In total, each session will be lasting approximately 45-60 minutes and a physiotherapist or personal trainer will supervise each session. Depending on the participants starting point, there will be 3 supervised session per week and two sessions where the participants do activity with low intensity (walk) by themselves and keep a log with duration (time) and intensity (using Borg scale).
  Interventions: Other: Physical activity
- Controls (No Intervention): These patients will be acting as controls by not been instructed to physical activity. We will not monitor their activity either as this has been shown to increase activity by itself.

INTERVENTIONS:
Other: Physical activity — Aerobic physical activity as stated in Arm A
  Arms: Physical aerobic intervention

SUMMARY:
Previous research into metabolic and hypoxic markers has found evidence of preclinical impact of exercise on prostate tumor blood flow and oxygenation in rodents . As radiotherapy is a frequently used and effective therapy for and that sufficient oxygenation is decisive to the effect of radiotherapy, an underlying hypothesis that aerobic exercise might improve treatment efficacy of radiotherapy in prostate cancer is put forward. This study has a potential challenging intervention, but a potential very high gain as it includes active patient participation to significantly improve outcome of radical radiotherapy.

DETAILED DESCRIPTION:
A randomized controlled trial with four to five weeks of moderate/high intensity aerobic exercise program compared with no intervention for 32 prostate cancer patients waiting for radical prostatectomy at the University Hospital of North Norway (UNN). 16 patients will undergo the intervention. The expression of the hypoxic marker pimonidazole in the prostate specimens of intervention groups and the control groups will be assessed. This method is considered a reliable tissue oxygenation measurement technique. These patients will also have their and blood flow and hypoxia measured in prostate cancers through magnetic resonance imaging (MRIs).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed PC
* planned radical prostatectomy
* informed consent given
* above 18 years of age
* BMI < 30
* non-smoker
* living in Tromso region

Exclusion Criteria:

* Contraindications to the intervention like;

  * heart failure,
  * angina pectoris,
  * respiratory disease limiting possible intervention
  * use of physical supportive devices to aid movement
* High level of physical activity
* smoking
* BMI>30

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Hypoxic fraction-gold standard | through study completion, an average of 1 year
  We will measure the hypoxic fraction in prostate cancer specimens by pimonidazole

SECONDARY OUTCOMES:
Side effects | through study completion, an average of 1 year
  We will use the Expanded Prostate Cancer Index Composite (EPIC) designed to evaluate patient function and side effects after PC treatment in both groups
Hypoxic fraction-MRI | through study completion, an average of 1 year
  We will try to explore the hypoxic fraction by use of magnetic resonance imaging
Health related Quality of life | through study completion, an average of 1 year
  We will use EORTC-QLQ30 which is a validated instrument designed to measure quality of life in prostate cancer in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Sigve Andersen, MD, PhD, Principal Investigator — UNN HF Tromsø
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No